CLINICAL TRIAL: NCT00774202
Title: A Rand. Trial Comp Higher Doses of Rituximab (Rituxan) With Standard Doses of Rituxan in Combination With CVP (Cyclophosphamide, Vincristine, and Prednisone) in Patients With Chronic ITP Who Have Failed/Relapsed After Rituxan Treatment
Brief Title: Higher Dose of Rituxan Versus Standard Doses of Rituxan With Cyclophosphamide, Vincristine, and Prednisone in Subjects With Chronic ITP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Biogen (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0301005964
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Pts w/ Chronic ITP who have fail/relap after Rituxan rx
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rituximab, Cyclophosphamide, Vincristine, Prednisone (Active Comparator): 'Standard Dose of Rituximab administered with C, V, P (CVP)'
  Interventions: Rituximab will be administered as an IV infusion at the standard dose of 375 mg/m2 for 4 doses at standard rates and use of premedication. The schedule will be to give the first rituximab infusion 5 days (± 3 days) prior to first administration of CVP, and the following 3 infusions will be given on the same day as the 3 cycles of C, V, P. On those days, the IV Cyclophosphamide and Vincristine will be given first so that the administration of fluids with the rituximab can be used as post-cyclophosphamide hydration, Cyclophosphamide dosing will be 750mg/m2 (maximum 2000mg), vincristine 1.4 mg/m2 (up to 1.6 mg), prednisone 100mg po daily for 5 days.
  Interventions: Drug: Rituxan, Cyclophosphamide, Vincristine, Prednisone
- Higher Dose of Rituximab (Active Comparator): In this arm, Rituximab will be administered at a dose of 750 mg/m2 once a week x 4 consecutive weeks (4 infusions in total). We will perform EKG monitor tracings before, during and after Rituxan infusions. This will be a single-lead tracing that will allow us to look at the Q-T interval.
  Interventions: Drug: Higher Dose of Rituximab

INTERVENTIONS:
Drug: Rituxan, Cyclophosphamide, Vincristine, Prednisone — 'Rituximab, Cyclophosphamide, Vincristine, Prednisone interventions are as follows: Rituximab will be administered as an IV infusion at the standard dose of 375 mg/m2 for 4 doses. However, the schedule of the infusions will be different than the usual one: Rather than administrating the 4 doses once weekly, the first infusion will be given 5 days (± 3 days) prior to the first infusions of C and V and oral P, and the following 3 rituximab infusions will be given on the same day as the 3 cycles of C, V, and P.
  Other Names: Rituximab
  Arms: Rituximab, Cyclophosphamide, Vincristine, Prednisone
Drug: Higher Dose of Rituximab — rituximab 750mg/m2 (twice the standard dose of 375mg/m2) will be given weekly for 4 weeks. Premedication and infusion rate escalation will be exactly the same as for standard dose rituximab. The additional dose will thus run at 400ml/hr.
  Arms: Higher Dose of Rituximab

SUMMARY:
This study is designed to compare the efficacy and safety of higher doses of Rituxan with a regimen combining standard doses of Rituxan + CVP in patients with chronic ITP who did not respond to or relapsed after standard doses of Rituxan. Patients eligible for this protocol will be stratified into two subgroups according to their initial response to Rituxan.

DETAILED DESCRIPTION:
The rationale for using chemotherapy in combination with Rituximab:

Since Rituximab is an anti-B cell therapy, in order to improve the rate of durable responses beyond the 32% (18 of 57) seen with Rituximab alone, it seems appropriate to combine it with a therapy that would also target T cells and/or macrophages. Our plan is therefore to combine Rituximab with a standard chemotherapy (CHOP)-like regimen as previously successfully tested in patients with follicular or diffuse large-B-cell lymphomas 13-15. The "CHOP" chemotherapy regimen is a combination of cyclophosphamide, doxorubicin, vincristine and prednisone (or prednisolone) that has been considered the "gold standard" for treating lymphomas for more than 20 years.

This combination of medications was used in a Hodgkin's patient with refractory ITP and became the template for developing the use of cyclophosphamide, vincristine, and prednisone for ITP as initially reported in 1993. Since reports on doxorubicin efficacy by itself in ITP are only anecdotal 16 and this drug has a potential cardiac toxicity, a CVP regimen (namely a combination of cyclophosphamide + vincristine and prednisone) should be similar in efficacy to CHOP in patients with ITP and have less toxicity. Indeed, the efficacy of such a chemotherapy12 as well as pulses cyclophosphamide therapy alone11 have already been reported in patients with refractory ITP.

Since attempts to increase the efficacy of CHOP by increasing the doses or adding other cytotoxic drugs have failed, a new therapeutic strategy combining CHOP with Rituxan has been successfully developed in the last few years in various types of B-cell lymphomas 13-15. In elderly patients with diffuse large-B-cell lymphoma, the addition of Rituxan to standard CHOP chemotherapy significantly reduced the risk of treatment failure and deaths without increasing toxicity 13. Moreover, in autoimmune disorders, there are few preliminary data suggesting that Rituxan and cyclophopshamide given in combination could be effective and relatively safe in patients with active rheumatoid arthritis 17.

Therefore, the rationale for combining Rituxan with a CHOP-like regimen in ITP is threefold:

Both Rituxan and CHOP or IV cyclophosphamide have efficacy in ITP The treatments have different mechanisms of action. They have minimally-overlapping toxicities.

The rationale for using higher doses of Rituxan in patients who had no response, or relapsed, to the drug at the standard dose:

The standard dose of Rituxan is arbitrary in that one dose of Rituxan has been used in the great majority of the clinical trials and virtually all patients since the FDA approval of Rituxan in 1997: 375 mg/m2 weekly x 4 weeks. To date, because Rituxan is a monoclonal antibody rather than a chemotherapeutic agent, it was recognized that a true maximum tolerated dose (MTD) might not be achieved. Among other factors that could influence the tolerance of higher doses of Rituxan are the rate of CD20 surface expression and the serum level of the antibody11. Limited trials of higher doses have been pursued in CLL18 (up to 2,250 mg/m2 per dose), but not in other types of lymphoma or in autoimmune diseases. In CLL, mild to severe toxicity was exclusively observed with the first dose (375 mg/m2) while toxicity on subsequent higher doses was minimal. In ITP, some of the few patients that have been retreated responded better to the second dose of rituximab than to the initial treatment (although the opposite is also true). Full depletion of the marrow and especially the lymph nodes is not achieved by the current dose regimen and B cells return in substantial number to the peripheral blood within 3-6 months in patients with ITP treated at the conventional dose. We therefore anticipate that in ITP patients who relapsed or did not respond after a previous course of rituximab, doubling the dose could lead to a deeper and more prolonged B cell depletion and to a better increase in the platelet count without enhancing toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to participate in the study if they:

* Have chronic ITP19 (> 6 months duration)
* Have received Rituximab a minimum of 3 months prior to entry
* Have received no more than 2 courses of Rituximab at standard dose separated by a minimum of 12 weeks
* Have not achieved a durable response to Rituximab, with platelet counts < 30,000/ml when not supported by other treatment
* Have a platelet count of < 30,000/ul on two separate occasions 1-2 weeks apart within the past month prior to the inclusion
* We will allow patients who do not have 2 platelet counts < 30,000 on two separate occasions 1-2 weeks apart in the past month, as long as they have either Evan's Syndrome or autoimmune neutropenia (have hemoglobin < 10 g/dL and reticulocytes > 4%, or an absolute neutrophil count < 1.0 K/uL twice within 1 month)
* Are age ≥ 10 years old
* Male and Female
* Had a splenectomy at least 60 days prior to study entry, or a contraindication to splenectomy
* Give written informed consent
* Use an effective means of contraception during treatment and for six months after completion of treatment
* Have negative serum pregnancy test, for all women who are able to have children, within 14 days prior to study entry

Exclusion Criteria:

Male and female subjects will be ineligible to participate if they:

* Received prior treatment with cyclophosphamide within the last 3 months
* Received prior treatment with > 4 infusions of vinca alkaloids within the 6 months
* Had previous or concomitant malignancy other than basal cell or squamous cell carcinoma of the skin, carcinoma-in-situ of the cervix, or other malignancy for which the patient had not been disease-free for at least 5 years
* Have a HIV infection
* Have hepatitis Bs antigen positivity or active hepatitis C infection
* Have an absolute neutrophil count < 1.000/mm3 at study entry (unless related to autoimmune neutropenia)
* Have a Hemoglobin level < 10 g/dl other than caused by thalassemia trait, iron deficiency or autoimmune hemolytic anemia (patients with Evan's syndrome will not be excluded)
* Have an impaired renal function as indicated by a serum creatinine level > 2.0 mg/dL
* Have an inadequate liver function as indicated by a total bilirubin level > 2.0 mg/dL and/or an AST or ALT level > 3x upper limit of normal
* Have active infection requiring antibiotic therapy within 7 days prior to study entry
* Are pregnant or lactating women, or plan to become pregnant or impregnated within 12 months of receiving study drug
* Have had a prior severe reaction to Rituximab, leading to discontinuation of treatment
* Have a New York Heart Classification III or IV heart disease
* Have a history of severe psychiatric disorder or are unable to comply with study and follow-up procedures

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Bussel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- 525 East 68th Street, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
publication of data in American journal of hematology
Time Frame: soon (2009)
Access Criteria: journal subscribers

REFERENCES:
- [Result] Hasan A, Michel M, Patel V, Stasi R, Cunningham-Rundles S, Leonard JP, Bussel J. Repeated courses of rituximab in chronic ITP: Three different regimens. Am J Hematol. 2009 Oct;84(10):661-5. doi: 10.1002/ajh.21512. PMID 19731307
- See also: http://onlinelibrary.wiley.com/doi/10.1002/ajh.21512/epdf — http://onlinelibrary.wiley.com/doi/10.1002/ajh.21512/abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose of Rituxan Plus CVP (R-CVP): 'Rituxan + Cyclophosphamide, Vincristine and Prednisone (R-CVP). Rituximab administered as an IV infusion at the standard dose of 375 mg/m2 for 4 doses. First Rituxan infusion will be given 5 days (± 3 days) prior to the first CVP, and the following 3 infusions will be given on the same day as the 3 cycles of CVP at week 2, week 5, and week 8.
- Double Dose of Rituximab: Rituximab administered at a dose of 750 mg/m2 once a week x 4 consecutive weeks (4 infusions in total).
Period: Overall Study
Arm/Group | Standard Dose of Rituxan Plus CVP (R-CVP) | Double Dose of Rituximab
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 17 patients total treated and analysis is of responding patients for efficacy and SAE for safety
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose of Rituxan Plus CVP (R-CVP) | Double Dose of Rituximab | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Customized [Mean (Standard Deviation); unit: years] — age > 12 years of age
  years
    age continuous | 36 (17) | 44 (19) | 40 (10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males entered at Baseline | 4 | 4 | 8
  Females entered at baseline | 5 | 4 | 9
Initial response to treatment with standard dose rituximab [Count of Participants; unit: Participants] — complete response (CR) is a stable platelet count > 100,000/uL on no ongoing treatment a partial response (PR) is a platelet count > 30,000/uL and doubling of baseline platelet count on no ongoing treatment that is not a CR non-response is neither a CR or a PR
  Participants
    Complete Response (CR) | 4 | 4 | 8
    Partial Response (PR) | 1 | 1 | 2
    No Response (NR) | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Higher Double Doses of Rituxan and of Standard Dose of Rituxan + Cyclophosphamide, Vincristine, Prednisone
Description: Outcome measure was determined by comparing the study participants' historical responses to their initial treatment of rituximab at standard dose/regimen without "enhancement" (based on duration of response and type of response) to the participants response to their study treatment responses. Thus each patient was his or her own control although all study treatments included standard dose rituximab treatments (one at double the dose and one with additional treatments).
Time Frame: 2 years
Population: the number of patients in each arm that increase their platelet count consistently above 100,000/uL after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dose of Rituxan Plus CVP (R-CVP) | Double Dose of Rituximab
Number analyzed (Participants) | 9 | 8
Participants
  same response as historical rituximab | 8 | 7
  Worse Response | 1 | 1
  Better Response | 0 | 0

2. Secondary Outcome: Number of Participants With SAEs
Description: How many participants had SAEs among those receiving R-CVP or among those receiving double dose rituximab and did participants in one arm have substantially more SAEs than those in the other arm
Time Frame: 2 years
Measure: Number; unit: number of patients with SAEs
Groups:
- Rituximab + CVP: patients receiving rituximab and cyclophosphamide and vincristine and prednisone
- Double Dose Rituximab: :patients receiving double dose rituximab
Arm/Group | Rituximab + CVP | Double Dose Rituximab
Number analyzed (Participants) | 9 | 8
number of patients with SAEs | 0 | 1

3. Secondary Outcome: Relative Efficacy of the 2 Groups
Description: The goal is to see if there are major differences between the two arms for each group in term of efficacy and of toxicity both overall and in comparison to the previous responses to rituximab alone. The comparisons are for level of response eg CR (>100k) vs PR (230-100k) vs NR (<30k) and for duration of response-----duration of response is controlled by comparison to duration of response from initial rituximab infusions
Time Frame: 2 years
Measure: Number; unit: number of responders
Groups:
- Rituximab, C, V, P: rituximab, cyclophosphamide, vincristine, prednisone
- High Dose Rituximab: double the dose of rituximab
Arm/Group | Rituximab, C, V, P | High Dose Rituximab
Number analyzed (Participants) | 9 | 8
number of responders
  CR | 4 | 4
  PR | 1 | 0
  response longer than previous response | 0 | 0

ADVERSE EVENTS:
Time Frame: collected over 2 years
Description: based on adverse event reporting
Arm/Group | Rituximab + C, V, P | Double Dose Rituximab
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8
Other Adverse Events (participants affected / at risk) | 4/9 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + C, V, P (N=9) | Double Dose Rituximab (N=8)
Serum Sickness (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + C, V, P (N=9) | Double Dose Rituximab (N=8)
non-serious (General disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes